CLINICAL TRIAL: NCT03165669
Title: Randomized, Controlled Clinical Trial With Cross-over on the Efficacy of Cervical Pillows and an Educational Intervention in Patients With Chronic Non-specific Neck Pain
Brief Title: Evaluation of the Efficacy of Cervical Pillows in Subjects With Non-specific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: SOFF-ART S.r.l. (Unknown)
Responsible Party: Principal Investigator, Paolo Pillastrini, Professore ordinario, University of Bologna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1202/2017
Record Dates: First submitted 2017-05-20; First posted 2017-05-24 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Neck Pain
Keywords: education; sleep; pillow; neck
MeSH Terms: conditions — Neck Pain | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Two groups of patients will be randomized in two parallel arms. At Time zero, the first one will receive education, the second one cervical pillow. After 4 weeks, the 1st follow-up will be done (Time one), and after 4 weeks of wash-out, the 2nd follow-up will be done (Time two). At this moment, the group that received cervical pillow will receive education, and vice versa. After 4 weeks (Time three), the final follow-up will be done.
  be done.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator will receive the results of outcome measures without any information of the group assignement.
  The outcome assessors will be masked on the group assignment, because they will receive only the list of participants,without the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical pillow (Experimental): The cervical pillow is known as the Viscospring PostuRite - "medium" model, made by SOFF-ART S.r.l. - Via Maestri del Lavoro 49 - 05100 Terni, Italy. The "Viscospring PostuRite" pillow is externally made of viscoelastic polyurethane and internally 60 independent, individually coated harmonic phosphate-coated steel springs, are thought to promote correct posture of the cervical spine, due to the adaptation of the pillow to the shape and movements of the head.
  Each intervention will be supported by a 30-minutes informative session delivered by a physical therapist, and will be completed by the delivery of an informative brochure.
  Interventions: Device: Viscospring PostuRite - "medium" model
- Education (Active Comparator): The educational intervention will be conducted by a physical therapist and will consist of a advice on positions, movements and activities recommended or not recommended for people with chronic neck pain, both in the workplace and in leisure time, including nighttime postures. Each educational intervention will be carried out individually, will last half an hour and will be supported by the delivery of an informative brochure.
  Interventions: Other: Education

INTERVENTIONS:
Device: Viscospring PostuRite - "medium" model — Cervical pillow use, 30-minutes instruction session supported by a brochure
  Other Names: Cervical pillow
  Arms: Cervical pillow
Other: Education — 30-minutes educational session delivered by a physical therapist and supported by an informative brochure.
  Arms: Education

SUMMARY:
This randomized controlled with cross-over trial aims to investigate the efficacy of a cervical pillow (the "Viscospring PostuRite" made by SOFF-ART S.r.l. Via Maestri del Lavoro 49 - 05100 Terni, Italy) versus education in non-specific chronic neck pain. More specifically, effectiveness will be measured using the following outcome measures: pain, disability, sleep quality, cervical pillow satisfaction, and global perception of the treatment effectiveness.

DETAILED DESCRIPTION:
The cervical pillow intervention will consist of the delivery and use of a particular cervical pillow ("Viscospring Postural") to be used during nighttime sleep. Each intervention will include an individual meeting with a physical therapist who will explain how to use and maintain the pillow, will last half an hour, and will be supported by the delivery of a user manual. There will be an opportunity to clarify any concerns and to receive answers to questions.

The educational intervention will be conducted by a physical therapist and will consist of advice on proper positions, movements, and activities recommended or not recommended for people with chronic neck pain, both in the workplace and in leisure time, including nighttime postures. Each educational intervention will be carried out individually, will last half an hour, and will be supported by the delivery of an informative brochure. There will be an opportunity to clarify any concerns and to receive answers to questions.

Participants will be required during the duration of the study refrain from modifying the dosage or type of prescribed analgesic or anti-inflammatory drugs they may be taking at the time the study starts and to refrain from initiating new drugs.

Participants will also be required refrain from undertaking any physical therapy or manipulative treatment for neck pain and to pursue their usual activities: work, recreation and physical activity.

Participants will also be required to complete a daily diary of pain for the duration of the study in order to monitor the development of any exclusion criterion during the period of study.

After the administration of the interventions (after 4 weeks of treatment - "Time one"), the first follow-up will be performed, with the administration of these questionnaires: Neck Disability Index (NDI-I), 0-100 Numerical Rating Scale, Pittsburg Sleep Quality Index (PSQI), Global Perceived Effect (GPE), Neck Pillow Satisfaction (NPS).

After four weeks from the " Time one" of the study, another follow-up will be performed, with the administration of the following questionnaires: Neck Disability Index (NDI-I), 0-100 Numerical Rating Scale, Pittsburg Sleep Quality Index (PSQI), and crossover will be performed, which consists in the exchange of treatments between the two groups: the group that did the first intervention will receive the second, and vice versa.

Four weeks after the cross-over, the third follow-up will be performed ("Time three"). In this final phase of the study, these questionnaires will be administrated: Neck Disability Index (NDI-I), 0-100 Numerical Rating Scale, Pittsburg Sleep Quality Index (PSQI), Global Perceived Effect (GPE), Neck Pillow Satisfaction (NPS).

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific chronic neck pain (neck pain from 3 months or more, not related to specific pathologies);
* Neck pain, with or without irradiation to the upper limb or to the head, noted as ≥2 on a scale of 0-10;
* Good comprehension of written and spoken Italian language;
* Informed consent.

Exclusion Criteria:

* Acute or sub-acute neck pain;
* Specific causes of cervical pain (trauma, herniated disc, vertebral deformity, fractures, dislocations);
* Central or peripheral neurological signs;
* Systemic pathologies;
* Rheumatic disorders;
* Neuromuscular pathologies;
* Tumors;
* Cognitive deficits;
* Surgical interventions in the last six months prior to the study;
* Physiotherapeutic treatments in the last six months prior to the study;
* To modify the type or the dosage of analgesic or anti-inflammatory drugs taken at baseline or new drug intakes;
* Using no pillow or 2 pillows during night time sleep.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in neck pain over time at 4, 8 and 12 weeks | At baseline, and at 3 follow-ups (after 4, 8, and 12 weeks)
  0-100 Numerical Rating Scale for neck, shoulders, thoracic pain, and headache. Frequency of neck, shoulders, thoracic pain, and headache.

SECONDARY OUTCOMES:
Changes in neck disability over time at 4, 8 and 12 weeks | At baseline, and at 3 follow-ups (after 4, 8, and 12 weeks)
  Neck Disability Index - Italian version
Changes in Global Perceived Effect (GPE) over time at 4 and 12 weeks | After 4 and 12 weeks from baseline
  One question on a 7 points Likert scale
Changes in Neck Pillow Satisfaction (NPS) over time at 4 and 12 weeks | After 4 and 12 weeks from baseline
  One question on a 7 points Likert scale
Changes in sleep quality over time at 4, 8 and 12 weeks | At baseline, and at 3 follow-ups (after 4, 8, and 12 weeks)
  Pittsburgh Sleep Quality Index - Italian version

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, Principal Investigator — University of Bologna
Locations (2):
- Italy (2):
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - University of Bologna, Bologna, Emilia-Romagna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro-Martin E, Ortiz-Comino L, Gallart-Aragon T, Esteban-Moreno B, Arroyo-Morales M, Galiano-Castillo N. Myofascial Induction Effects on Neck-Shoulder Pain in Breast Cancer Survivors: Randomized, Single-Blind, Placebo-Controlled Crossover Design. Arch Phys Med Rehabil. 2017 May;98(5):832-840. doi: 10.1016/j.apmr.2016.11.019. Epub 2016 Dec 18. PMID 28003133
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333
- [Background] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760
- [Background] Domingo AR, Diek M, Goble KM, Maluf KS, Goble DJ, Baweja HS. Short-duration therapeutic massage reduces postural upper trapezius muscle activity. Neuroreport. 2017 Jan 18;28(2):108-110. doi: 10.1097/WNR.0000000000000718. PMID 27977513
- [Background] Erfanian P, Tenzif S, Guerriero RC. Assessing effects of a semi-customized experimental cervical pillow on symptomatic adults with chronic neck pain with and without headache. J Can Chiropr Assoc. 2004 Mar;48(1):20-8. PMID 17549216
- [Background] Gordon SJ, Grimmer-Somers K, Trott P. Pillow use: the behaviour of cervical pain, sleep quality and pillow comfort in side sleepers. Man Ther. 2009 Dec;14(6):671-8. doi: 10.1016/j.math.2009.02.006. Epub 2009 May 7. PMID 19427257
- [Background] Hagino C, Boscariol J, Dover L, Letendre R, Wicks M. Before/after study to determine the effectiveness of the align-right cylindrical cervical pillow in reducing chronic neck pain severity. J Manipulative Physiol Ther. 1998 Feb;21(2):89-93. PMID 9502063
- [Background] Haines T, Gross AR, Burnie S, Goldsmith CH, Perry L, Graham N; Cervical Overview Group (COG). A Cochrane review of patient education for neck pain. Spine J. 2009 Oct;9(10):859-71. doi: 10.1016/j.spinee.2009.04.019. Epub 2009 Jul 12. PMID 19596214
- [Background] Helewa A, Goldsmith CH, Smythe HA, Lee P, Obright K, Stitt L. Effect of therapeutic exercise and sleeping neck support on patients with chronic neck pain: a randomized clinical trial. J Rheumatol. 2007 Jan;34(1):151-8. PMID 17216683
- [Background] Lavin RA, Pappagallo M, Kuhlemeier KV. Cervical pain: a comparison of three pillows. Arch Phys Med Rehabil. 1997 Feb;78(2):193-8. doi: 10.1016/s0003-9993(97)90263-x. PMID 9041902
- [Background] Monticone M, Ferrante S, Vernon H, Rocca B, Dal Farra F, Foti C. Development of the Italian Version of the Neck Disability Index: cross-cultural adaptation, factor analysis, reliability, validity, and sensitivity to change. Spine (Phila Pa 1976). 2012 Aug 1;37(17):E1038-44. doi: 10.1097/BRS.0b013e3182579795. PMID 22487712
- [Background] Klaber Moffett JA, Jackson DA, Richmond S, Hahn S, Coulton S, Farrin A, Manca A, Torgerson DJ. Randomised trial of a brief physiotherapy intervention compared with usual physiotherapy for neck pain patients: outcomes and patients' preference. BMJ. 2005 Jan 8;330(7482):75. doi: 10.1136/bmj.38286.493206.82. Epub 2004 Dec 7. PMID 15585539
- [Background] Persson L, Moritz U. Neck support pillows: a comparative study. J Manipulative Physiol Ther. 1998 May;21(4):237-40. PMID 9608378
- [Background] Sacco IC, Pereira IL, Dinato RC, Silva VC, Friso B, Viterbo SF. The effect of pillow height on muscle activity of the neck and mid-upper back and patient perception of comfort. J Manipulative Physiol Ther. 2015 Jul-Aug;38(6):375-81. doi: 10.1016/j.jmpt.2015.06.012. Epub 2015 Jul 21. PMID 26209581
- [Background] Wegner S, Jull G, O'Leary S, Johnston V. The effect of a scapular postural correction strategy on trapezius activity in patients with neck pain. Man Ther. 2010 Dec;15(6):562-6. doi: 10.1016/j.math.2010.06.006. Epub 2010 Jul 21. PMID 20663706
- [Background] Young BA, Walker MJ, Strunce JB, Boyles RE, Whitman JM, Childs JD. Responsiveness of the Neck Disability Index in patients with mechanical neck disorders. Spine J. 2009 Oct;9(10):802-8. doi: 10.1016/j.spinee.2009.06.002. Epub 2009 Jul 25. PMID 19632904
- [Derived] Vanti C, Banchelli F, Marino C, Puccetti A, Guccione AA, Pillastrini P. Effectiveness of a "Spring Pillow" Versus Education in Chronic Nonspecific Neck Pain: A Randomized Controlled Trial. Phys Ther. 2019 Sep 1;99(9):1177-1188. doi: 10.1093/ptj/pzz056. PMID 30939188